CLINICAL TRIAL: NCT03665298
Title: Needle-X: Usability Testing of a Smartphone Application
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never started by the responsible party (medical student who is no longer at the institution).
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-00652
Record Dates: First submitted 2018-08-14; First posted 2018-09-11 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Needle X (Experimental): Smartphone application application to enhance access to sterile needles, naloxone overdose kits, and addiction treatment programs in New York City.
  Interventions: Behavioral: Smartphone Application

INTERVENTIONS:
Behavioral: Smartphone Application — App that helps patients find syringe exchange programs, safe way to dispose of needles, access to naloxone kits and access to free medical care and addiction treatment programs.

SUMMARY:
Mobile health interventions offer a longitudinal approach to reducing the burden of substance use disorders and may stem the rise of the opioid overdose epidemic. Smartphone applications are one of the most popular mobile phone features nationally, among patients in addiction treatment, and among criminal justice involved (CJI) patients enrolled in addiction treatment. This research conducted at Bellevue Hospital's inpatient detoxification program established attitudes and self-reported behaviors favorable to theoretical smartphone applications addressing opioid use, HIV, and HCV prevention and management strategies. This study aims to assess the feasibility and usability of a smartphone application to enhance access to sterile needles, naloxone overdose kits, and addiction treatment programs in New York City.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in spoken and written English;
* Meets or has previously met DSM-5 criteria for current opioid use disorder, of at least moderate severity;
* Owns or has owned a smartphone

Exclusion Criteria:

* Any patient who does not meet the inclusion criteria as above, is clinically unstable per the unit admitting physicians, refuses to participate in the study, or is cognitively impaired.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Needle-X application | 12 Months
  number of patients enrolled, as this study will include a single interaction, at which point the patient will no longer be part of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Babak Tofighi, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Violates the ethical conduct of technology based intervention research for an early-stage intervention development project.